CLINICAL TRIAL: NCT07161089
Title: Correlation Between Knowledge, Attitudes and Practices of Caregivers and Oral Health Status of Alzheimer's Disease Patients in Cairo: A Cross-Sectional Study
Brief Title: Correlation Between Knowledge, Attitude and Practices of Caregivers and Oral Health Status of Alzheimer's Disease Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherine Tarek Mohamed Elsayed Khaled, Principal investigator, Cairo University
Other Study IDs: CU 25 8 2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Practices of Caregivers; Knowledge of Caregivers; Attitudes of Caregivers; Oral Health Status of Alzheimer Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- caregivers of Alzheimer's disease patients: knowledge, attitudes and practices of primary caregivers of Alzheimer's disease patients
- Alzheimer's disease patients: oral health status of Alzheimer's disease patients

SUMMARY:
A cross-sectional study to assess the relation between the knowledge, attitude and practices or caregivers of Alzheimer's disease patients and the oral health status of these patients.

DETAILED DESCRIPTION:
A cross-sectional study to assess knowledge, attitude and practices of care givers of Alzheimer's disease patients using a questionnaire as a tool and evaluating the oral health status of these patients by recording DMF scores and simplified oral hygiene index in order to assess if there is any correlation between those two variables

ELIGIBILITY:
Inclusion Criteria for caregivers:

* all primary caregivers serving Alzheimer's disease patients.

Inclusion criteria for Alzheimer's disease patients :

* all patients whose medical condition allows for an oral examination

Exclusion Criteria for caregivers:

* caregivers who are not directly involved in the daily care
* caregivers who refuse to participate in the study

Exclusion criteria for Alzheimer's disease patients :

* patients with deteriorated medical condition that do not permit clinical examination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: for caregivers: all employed caregivers in the center involved. in the care of Alzheimer's disease patients .
  for Alzehimer's disease patients: all Alzheimier's disease patients residing in the center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
knowledge , attitude and practices of primary caregivers of Alzheimer's disease patients | Baseline
  validated questionnaire to assess the KAP of caregivers of AD patients

SECONDARY OUTCOMES:
Oral health status of AD patients | Baseline
  measure the DMF index

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided